CLINICAL TRIAL: NCT06598722
Title: The Efficacy and Safety of BCL-2 Inhibitors Combined with the HyperCVAD Regimen in the Treatment of Newly Diagnosed T-lymphoblastic Leukemia/ Lymphoma
Brief Title: BCL-2 Inhibitors Combined with the HyperCVAD Regimen for Newly Diagnosed T-lymphoblastic Leukemia/lymphoma.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Investigator Official Title, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-T-LBL-VEN-2024
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Lymphoblastic Lymphoma, Adult; Lymphoblastic Leukemia, Acute T-cell
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCL-2 inhibitors combined with the HyperCVAD regimen for newly diagnosed T-ALL/LBL (Experimental)
  Interventions: Drug: BCL-2 inhibitors combined with the HyperCVAD regimen
- propensity score matching with historical data (Other)
  Interventions: Other: Propensity score matching historical data

INTERVENTIONS:
Drug: BCL-2 inhibitors combined with the HyperCVAD regimen — BCL-2 inhibitors combined with the HyperCVAD regimen for newly diagnosed adult T-ALL/LBL
  Arms: BCL-2 inhibitors combined with the HyperCVAD regimen for newly diagnosed T-ALL/LBL
Other: Propensity score matching historical data — Propensity score matching was conducted with historical data (matching factors included age, gender, initial LDH levels, and the presence or absence of a large mediastinal mass at diagnosis) to compare the advantages and disadvantages of the experimental regimen with previous induction treatment protocols.
  Arms: propensity score matching with historical data

SUMMARY:
The experimental group included patients diagnosed with T-ALL/LBL (T-lymphoblastic leukemia/ lymphoma) at initial diagnosis, who received treatment with BCL-2 inhibitors combined with the Hyper CVAD regimen. The control group consisted of patients diagnosed with T-ALL/LBL from multiple centers, for whom basic information, disease information, treatment details, and efficacy data were collected. Propensity score matching was conducted with historical data (matching factors included age, gender, initial LDH levels, and the presence or absence of a large mediastinal mass at diagnosis) to compare the advantages and disadvantages of the experimental regimen with previous induction treatment protocols. The primary endpoint was the complete remission (CR) rate after induction chemotherapy, while secondary endpoints included duration of remission (DOR), progression-free survival (PFS), overall survival (OS), and the occurrence of adverse events. This study aims to provide a more effective and safer treatment option for patients with T-LBL.

ELIGIBILITY:
Inclusion Criteria Age 18-60 years, regardless of gender; Expected survival time greater than 12 weeks; ECOG score 0-2; Pathologically or flow cytometrically confirmed as T-cell lymphoblastic lymphoma, with less than 25% tumor cell proportion in bone marrow smears;

Liver and kidney function, as well as cardiopulmonary function, meet the following requirements:

Creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 mL/min; Left ventricular ejection fraction greater than 50%, with no clinically significant ECG changes; Baseline oxygen saturation greater than 92% Total bilirubin ≤1.5×ULN; ALT and AST ≤3×ULN Able to understand the trial and has signed the informed consent form Exclusion Criteria A history of acute T-cell leukemia, T-cell lymphoma, or T-cell lymphoblastic lymphoma within the past 5 years, except for adequately treated carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin, localized prostate cancer after radical surgery, ductal carcinoma in situ after radical surgery, or thyroid cancer after radical surgery Active bacterial, viral, or fungal infections that require treatment and are not controlled; those who are HBsAg or HBcAb positive, with peripheral blood HBV DNA ≥ the lower limit of detection; individuals who are positive for hepatitis C virus antibodies and have positive peripheral blood HCV RNA; individuals who test positive for syphilis (TRUST test); individuals who are positive for human immunodeficiency virus (HIV) antibodies Dysfunction of important organs (cardiovascular, pulmonary) or a history of active gastrointestinal bleeding within the past 3 months; individuals with uncontrolled hypertension, hypertensive crisis, or a history of hypertensive encephalopathy, and a history or evidence of significant cardiovascular risk, including any of the following: congestive heart failure, unstable angina, clinically significant arrhythmias (e.g., ventricular fibrillation, ventricular tachycardia); a history of arterial thrombosis within the past 3 months (e.g., stroke, transient ischemic attack); a history of symptomatic deep vein thrombosis, pulmonary embolism within the past 6 months, or a history of coronary angioplasty, defibrillation, or any clinical complications or diseases that may pose a risk to the participant's safety or interfere with the evaluation, procedures, or completion of the study Any uncontrolled active disease that may interfere with participation in the trial; Active, uncontrolled central nervous system diseases or a history of central nervous system disease requiring treatment (e.g., epilepsy) Pregnant or breastfeeding women; and individuals planning to become pregnant within 1 year after infusion, during treatment, or after treatment ends Presence of uncontrolled active infections (except for simple urinary tract infections or upper respiratory infections Known allergies to any components of cyclophosphamide, doxorubicin, vincristine, cytarabine, methotrexate, etc.

Any situation that the investigator believes would compromise participant safety or interfere with the study objectives, or any individual deemed inappropriate for participation by the investigator Individuals with diseases affecting their ability to sign the written informed consent form or comply with study procedures; those unwilling or unable to adhere to study requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 206 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-08-07 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
AE | at the end of cycle 2(each cycle is 28 days)
  adverse events during research
The best overall response rate | at the end of cycle 2（each cycle is 28 days）
  complete remission and partial remission
Evaluate the best complete remission rate (CR) | at the end of cycle 4 of chemotherapy（each cycle is 28 days）

SECONDARY OUTCOMES:
Duration of remission | 1 year
  Duration of remission
OS | 1 year
  1 year overall survival
OS | 2 year
  2 year overall survival
PFS | 1 year
  1 year progression free survival
PFS | 2 year
  2 year progression free survival
the proportion of successful bridging to allogeneic hematopoietic stem cell transplantation | the end of the study
  he proportion of successful bridging to allogeneic hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided